CLINICAL TRIAL: NCT04170452
Title: HBV DNA Replication in Hepatocytes in HBV and HDV Co-infection
Brief Title: Study the Content of the HBV DNA in Liver Biopsy in the Patients Chronic Hepatitis Delta
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tokhirbek Dolimov (Other Government)
Responsible Party: Sponsor-Investigator, Tokhirbek Dolimov, Research Institute of Epidemiology, Microbiology and Infectious deseases, Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan
Organization: Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan (Other Government)
Other Study IDs: ADCC - 15.21.1
Record Dates: First submitted 2019-11-15; First posted 2019-11-20 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Chronic Hepatitis Delta; Liver Biopsy
Keywords: Viral hepatitis B; HBV DNA; Viral hepatitis Delta; iver biopsy; PCR
MeSH Terms: conditions — Hepatitis D, Chronic; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Detection of DNA HBV in liver cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Hepatitis Delta patients: Patients infected with delta virus
  Interventions: Procedure: liver biopsy

INTERVENTIONS:
Procedure: liver biopsy — Pre-procedure assessment of the liver with ultrasound should be performed for planning positioning and needle entrance point. Supine, oblique, or total left lateral decubitus are the possible positioning of the patient - it is important to make sure that the patient is comfortable and can remain still in that position. Assessing if the procedure will be performed under breath held and practice this with the patient. Marking of the entrance point on the skin is advised to aid the skin cleaning and dressing. A time-out should be performed by this stage. Skin site is prepped and draped to ensure asepsis. Ocal anaesthesia is infiltrated under the skin abdominal wall/intercostal space until the liver capsule. Entrance point is created with a scalpel. Using the freehand technique the needle is advanced under ultrasound guidance during the entire course of the biopsy. The needle tip must always cross the capsule prior to deploying the cutting device.

SUMMARY:
Study the content of the HBV DNA in liver biopsy in the patients with the Chronic Hepatitis Delta in absence of the HBV DNA in the blood plasma

DETAILED DESCRIPTION:
Investigators interpreted the data of several researchers that studied suppression of the HBV DNA replication in the Delta infection within this article. Co-infection and superinfection of hepatitis B virus (HBV) with hepatitis delta virus (HDV) leads to suppression of HBV replication in both patients as well as animals and cell models. The mechanisms underlying this suppression were not fully studied before.

Jaw-Ching Wu et al. described the suppression of HBV DNA replication during HBV and HDV co-infection for the first time in 1991. The results of studies in the liver experimental models HuH-7 clearly demonstrated that one delta HDV antigen can suppress the expression of HBV RNA.

Dulce Alfaiate et al. conducted studies on the experimental models proving that HBV replication markers, including HBeAg, total HBV DNA and pregenomic RNA were significantly reduced after superinfection with HDV which confirming the effect of HDV on HBV. But thereby, the levels of circularly covalently closed levels of HBV DNA (cccDNA) and HBsAg were not decreased. At the peak of HDV-RNA accumulation and appearance of the interference in HBV replication, a strong I type IFN response was observed with highly induced genes stimulated by the interferon, RSAD2 (Viperin) and IFI78 (MxA). Both mono- and superinfected dHepaRG cells maintained strong intracellular replication of HDV, which was accompanied with the strong secretion of infectious HDV virions.

The following analysis of the data in the experimental studies by Zhenfeng Zhang et al. proved that the HDV virus activated strongly IFN-β and IFN-λ in the hepatocyte cell lines. The active HDV replication induces the IFN-β/λ response. Unlike hepatitis B virus, hepatitis D virus infection causes a strong IFN-β/λ response in the innate immunocompetent cell lines. The activated IFN did not suppress replication of hepatitis D virus in vitro, which indicatesthat Delta hepatitis virus is resistant to the self-induced innate immune responses and therapeutic treatment for IFN.

According to the authors, this stimulation of the synthesis of endogenous IFN-β and IFN-λ inside the hepatocyte by the HDV virus caused suppression of the HBV virus replication.

The following study, conducted Paolo Pugnale et al., in Huh-7 human hepatoma cells demonstrates that HDV can disrupt the IFN-α-stimulated JAK-STAT signaling pathway (a mediating protein ensuring cell response to the signals from the interleukin receptors and growth factors). The mechanism adopted by HDV to interfere with IFN-α/β signaling is based on inhibition of the tyrosine phosphorylation of STAT1, STAT2 and Tyk2 receptor-bound kinase without reducing expression levels of the IFN receptor subunits or other components in the signaling cascade. These results indicate that the HDV virus develops a strategy to counteract the actions of I type IFN. This study may be useful for a better understanding of the observed resistance to IFN in the chronic patients with the Chronic Hepatitis Delta and may provide the useful data for defining new strategies for antiviral intervention.

However, it should be noted that KatashibaY. in his research indicates that IFN is mainly stimulated in case of infection with the DNA-containing viruses, while IL-12 induction predominates in case of the RNA-containing infections. Since HDV consists of a single-stranded RNA molecule, it is not expected to stimulate IFN.

Given the above stated disagreements in the results of the authors' studies, Investigators decided to examine the patients with the Chronic Hepatitis Delta when the HBV DNA was not detected in the blood during examination by PCR.

ELIGIBILITY:
Inclusion Criteria:

* patients with the Chronic Hepatitis Delta in absence of the HBV DNA in the blood plasma

Exclusion Criteria:

* patient's with the Chronic Hepatitis Delta in absence of the HBV DNA in the blood plasma but: inability to remain still and to maintain brief expiration for the procedure, suspected vascular lesion (eg, hemangioma), bleeding tendency (eg, INR > 1.2 despite receiving vitamin K, bleeding time > 10 min), severe thrombocytopenia (< 50,000/mL)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients with chronic viral hepatitis delta
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
The study the content of the HBV DNA in liver biopsy | up to 3 months
  In this study we are going to do liver biopsy in 30 patients with a diagnosis of Chronic Viral Hepatitis B and Delta.

CONTACTS AND LOCATIONS:
Overall Officials: Nariman Gulyamov, DSci, Study Chair — Research institute of epidemiology, microbiology and infectious diseases
Locations (1):
- RIEMID, Tashkent, Uchtepa District,, Uzbekistan

IPD SHARING:
Plan to Share IPD: No